CLINICAL TRIAL: NCT03241524
Title: Consistency of Three Different Questionnaires to Evaluating Sexual Functions in Young Healthy Women Before and After a Pelvic Floor Muscle Training Program
Brief Title: Consistency of Questionnaires to Evaluating Sexual Functions in Young Healthy Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Christiane Kelen Lucena da Costa, Graduate student, Universidade Federal do Rio Grande do Norte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 28032017
Record Dates: First submitted 2017-03-29; First posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Physical Activity
Keywords: Pelvic Floor muscles; Physical Therapy; Sexual function evaluation
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Sexual Dysfunctions, Psychological; Motor Activity

STUDY DESIGN:
Intervention Model Description: Perineal floor muscle performance and participants' sexual functions were evaluated in three successive situations: (1) Initial evaluation; (2) after 4 weeks (intermediate evaluation), and (3) 8 weeks (final evaluation) from the start of the training program.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (1):
- Exercise program for pelvic muscle floor (Experimental): Training program for pelvic muscles and application of 3 questionnaires for sexual function evaluation and the use of PERFECT and Perina methods to evaluate perineal musculature.
  Interventions: Other: Exercise program for pelvic muscle floor

INTERVENTIONS:
Other: Exercise program for pelvic muscle floor — Pelvic muscles of each participant was evaluated by PERFECT and Peritron methods in terms of strengthening as well as sexual function response using 3 questionnaires, before and after 4 and 8 weeks from the beggining of an exercise program prescribed according to individual ratings obtained in the previous evaluation.

SUMMARY:
The sample comprised 31 female undergraduate students attending a private University in João Pessoa, northeastern Brazil. The inclusion criteria were: age between 19 and 35 years, heterosexual, active sex life, living in a stable relationship for at least 6 months no pregnancy or parturition in the last 6 months, clinically healthy and agreeing with the terms for participating in the study. All participants gave their informed consent to take part in the study.

DETAILED DESCRIPTION:
PURPOSE: To compare the consistency of 3 instruments for sexual function evaluation in healthy young women before and after a pelvic floor muscle training. Methods: Thirty-one healthy young women were enrolled in an 8-week training program, consisting of bipedal exercises performed at home. The PERFECT and Peritron methods were used to estimate the efficacy of the intervention on pelvic muscles. Three questionnaires (FSFI, SQ-F and GRISS) were applied to assess sexual function. Both procedures were performed on three occasions: before, 4 and 8 weeks after the start of the training program. ANOVA for repeat measures and Tukey's post hoc were applied to analyze PERFECT and Peritron results, as well as individual domains and total scores of the questionnaires. The accuracy measured by the area under the ROC curve (AUC) for individual domains of each questionnaire and cross-validated pairwise comparison of the three instruments were also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age between 19 and 35 years;
* heterosexual with active sex life, living in a stable relationship for at least 6 months;
* no pregnancy or parturition in the last 6 months;
* clinically healthy;
* agreeing with the terms for participating in the study;
* To sign and agree with their informed consent to take part in the study.

Exclusion Criteria:

- Do not continue with the intervention program.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-03-12 (Actual); Primary Completion 2016-06-20 (Actual); Study Completion 2016-09-12 (Actual)

PRIMARY OUTCOMES:
Assessment of female sexual response by Female Sexual Function Inventory (FSFI) | 8 weeks
  This questionnaire contains 19 itens assessing sexual function over the past four weeks, associated with six domains and possible types of disorders: desire, arousal, lubrification, orgasm, satisfaction of sexual life, and pain during or after the intercourse.
Assessment of female sexual response by Sexual quotient for women (QS-F) | 8 weeks
  This instrument is composed of 10 questions that assess sexual function, adressing desire and interest in sex, foreplay, sexual arousal and harmony with the partner, comfort in sexual intercourse, and orgasm and sexual satisfaction. The overall scores range from 0 to 100, where high scores mean excellent sexual performance.
Assessment of female sexual response by Golombok-Rust Inventory of Sexual Satisfaction (GRISS) for female. | 8 weeks
  The GRISS is a 28-item questionnaire that provides a total GRISS score as well as two separate scales for males and females. For females, the scale has 8 items, including anorgasmia, vaginismus, non-communication, infrequency, female avoidance, female non-sensuality, female dissatisfaction and anorgasmia. Scoring was from 0 to 10 with values higher than 5 indicating sexual dysfunction.

SECONDARY OUTCOMES:
Pelvic floor muscles performance quantified by PERFECT method | 8 weeks
  This method is an acronym for the evaluation of contractile components of the pelvic floor muscles and was validated with high test-retest reliability, producing significant correlations for the variables, in particular, power and endurance. According to definitions of these methods, P indicates power or pressure, which corresponds to muscle strength estimated by manometry biofeedback or digital touch during voluntary maximum contraction. The evaluation is based on Oxford modified scale: Degrees: 0 - no perineal contraction visible or by palpation (non-contraction); 1- no perineal contraction visible, recognized only by palpation; 2 - weak perineal contraction to palpation; 3 - perineal contraction present, but with nonresistance to palpation; 4 - perineal contraction present with counter-resistance to palpation of less than 5 seconds ; and 5 - perineal contraction present with counter-resistance to palpation of more than 5 seconds.
Pelvic floor muscles performance quantified by PERITRON method | 8 weeks
  The Peritron is a hand-held clinical biofeedback perineometer used for assessing the strength of the pelvic floor muscles. The device helps teach patients how to effectively perform pelvic floor exercises (kegels). Pelvic floor contraction causes air pressure in the sensor to be transferred through the connecting tube and displayed on the readout unit.

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Physical Therapy, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sacomori C, Virtuoso JF, Kruger AP, Cardoso FL. [Pelvic floor muscle strength and sexual function in women]. Fisioterapia e Movimento, 28, 657-665, 2015.
- [Result] Damjanovic A, Duisin D, Barisic J. The evolution of the female sexual response concept: treatment implications. Srp Arh Celok Lek. 2013 Mar-Apr;141(3-4):268-74. doi: 10.2298/sarh1304268d. PMID 23745356
- [Derived] da Costa CKL, Spyrides MHC, de Sousa MBC. Consistency of three different questionnaires for evaluating sexual function in healthy young women. BMC Womens Health. 2018 Dec 20;18(1):204. doi: 10.1186/s12905-018-0693-y. PMID 30572853